CLINICAL TRIAL: NCT01163994
Title: Comparison of Ceftriaxone and Doxycycline for Treatment of Multiple Erythema Migrans
Brief Title: Antibiotic Treatment of Multiple Erythema Migrans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Franc Strle, M.D., PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEM-0510
Record Dates: First submitted 2010-07-13; First posted 2010-07-16 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Multiple Erythema Migrans
Keywords: erythema migrans; Lyme borreliosis; ceftriaxone treatment; doxycycline treatment; outcome; subjective symptoms
MeSH Terms: conditions — Glossitis, Benign Migratory; Lyme Disease | interventions — Ceftriaxone; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MEM-ceftriaxone (Active Comparator)
  Interventions: Drug: ceftriaxone
- MEM-doxycycline (Active Comparator)
  Interventions: Drug: doxycycline
- controls (No Intervention)
- EM-doxycycline (Active Comparator)
  Interventions: Other: erythema migrans patients treated with doxycycline

INTERVENTIONS:
Drug: ceftriaxone — intravenously, 2 g, qd, 15 days
  Arms: MEM-ceftriaxone
Drug: doxycycline — orally, 100 mg, bid, 15 days
  Arms: MEM-doxycycline
Other: erythema migrans patients treated with doxycycline — orally, 100 mg, bid, 15 days
  Arms: EM-doxycycline

SUMMARY:
The purpose of this study is to compare the efficacy and safety of 15-day ceftriaxone versus 15-day doxycycline treatment in patients with multiple erythema migrans.

ELIGIBILITY:
Inclusion Criteria:

* multiple erythema migrans in patients > 15 years

Exclusion Criteria:

* a history of Lyme borreliosis in the past
* pregnancy or lactation
* immunocompromised status
* serious adverse event to doxycycline or beta lactam antibiotic
* taking antibiotic with antiborrelial activity within 10 days

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2010-06; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Objective sequelae and post-treatment subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, dizziness, or irritability in patients treated for multiple erythema migrans with ceftriaxone or doxycycline for 15 days. | enrolling 3 years, 1 year follow-up for individual participant: first assessment at baseline
Objective sequelae and post-treatment subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, dizziness, or irritability in patients treated for multiple erythema migrans with ceftriaxone or doxycycline for 15 days. | second assessment at 14 days postenrollment
Objective sequelae and post-treatment subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, dizziness, or irritability in patients treated for multiple erythema migrans with ceftriaxone or doxycycline for 15 days. | third assessment at 2 months postenrollment
Objective sequelae and post-treatment subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, dizziness, or irritability in patients treated for multiple erythema migrans with ceftriaxone or doxycycline for 15 days. | fourth assessment at 6 months postenrollment
Objective sequelae and post-treatment subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, dizziness, or irritability in patients treated for multiple erythema migrans with ceftriaxone or doxycycline for 15 days. | fifth assessment at 12 months postenrollment

SECONDARY OUTCOMES:
Comparison of subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, or irritability between patients treated with antibiotic for multiple erythema migrans and control subjects without a history of Lyme borreliosis. | enrolling 3 years, 1 year follow-up for individual participant: first assessment at baseline
Objective sequelae and post-treatment subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, dizziness, or irritability in patients with solitary versus multiple erythema migrans after antibiotic treatment. | enrolling 3 years, 1 year follow-up for individual participant: at baseline and at 14 days, 2, 6, and 12 months thereafter
Comparison of subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, or irritability between patients treated with antibiotic for multiple erythema migrans and control subjects without a history of Lyme borreliosis. | second assessment at 6 months postenrollment
Comparison of subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, or irritability between patients treated with antibiotic for multiple erythema migrans and control subjects without a history of Lyme borreliosis. | third assessment at 6 months postenrollment
Objective sequelae and post-treatment subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, dizziness, or irritability in patients with solitary versus multiple erythema migrans after antibiotic treatment. | second assessment at 14 days postenrollment
Objective sequelae and post-treatment subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, dizziness, or irritability in patients with solitary versus multiple erythema migrans after antibiotic treatment. | third assessment at 2 months postenrollment
Objective sequelae and post-treatment subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, dizziness, or irritability in patients with solitary versus multiple erythema migrans after antibiotic treatment. | fourth assessment at 6 months postenrollment
Objective sequelae and post-treatment subjective symptoms such as fatigue, malaise, arthralgias, headache, myalgias, paresthesias, dizziness, or irritability in patients with solitary versus multiple erythema migrans after antibiotic treatment. | fifth assessment at 12 months postenrollment

CONTACTS AND LOCATIONS:
Overall Officials: Franc Strle, MD, Study Chair — UMC Ljubljana; Dasa Stupica, MD, Principal Investigator — UMC Ljubljana, Department of Infectious Diseases Ljubljana, Slovenia
Locations (1):
- UMC Ljubljana, Department of Infectious Diseases, Ljubljana, Slovenia

REFERENCES:
- [Derived] Veluscek M, Bajrovic FF, Strle F, Stupica D. Doxycycline-induced photosensitivity in patients treated for erythema migrans. BMC Infect Dis. 2018 Aug 3;18(1):365. doi: 10.1186/s12879-018-3270-y. PMID 30075748
- [Derived] Stupica D, Veluscek M, Blagus R, Bogovic P, Rojko T, Cerar T, Strle F. Oral doxycycline versus intravenous ceftriaxone for treatment of multiple erythema migrans: an open-label alternate-treatment observational trial. J Antimicrob Chemother. 2018 May 1;73(5):1352-1358. doi: 10.1093/jac/dkx534. PMID 29385444